CLINICAL TRIAL: NCT02397200
Title: Double Blind, Randomized , Placebo Controlled Study to Evaluate the Effect of Nutritional Supplementation on Growth of Short and Lean Adolescents Girls
Brief Title: Evaluating the Effect of Nutritional Supplementation on Growth of Short and Lean Adolescents Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: rmc000214ctil
Record Dates: First submitted 2015-02-24; First posted 2015-03-24 (Estimated); Last update posted 2025-05-16 (Actual); Status verified 2024-03

CONDITIONS: Growth Problem; Low Weight
Keywords: Growth; low weight; low height; Nutritional Supplementation
MeSH Terms: conditions — Thinness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional supplementation standardized formula (Experimental): Powder added to water, containing about 25% of recommended DRI for Calories, high protein (25% of calories) and multi vitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake )
  Interventions: Dietary Supplement: Nutritional supplementation standardized formula
- Placebo comparator (Placebo Comparator): Low caloric formula (Powder added to water), without added vitamins and minerals.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional supplementation standardized formula — Powder added to water, containing about 25% of recommended Daily Recommended Intake (DRI) for Calories, high protein (25% of calories) and multi vitamin and mineral (25%-100% of DRI for recommended daily allowance (RDA) or adequate intake )
  Arms: Nutritional supplementation standardized formula
Dietary Supplement: Placebo — Low caloric formula (Powder added to water), without added vitamins and minerals
  Arms: Placebo comparator

SUMMARY:
Study design:

Double blind, randomized, placebo controlled study. Participants will be randomly assigned either to the intervention group or the placebo control group. Randomization for the two study groups will be made in a ratio of 1:1.

The primary objective of the study is to assess the effect of 6-12 months treatment with nutritional supplementation standardized formula, in short and lean female adolescents on weight Standard Deviation Score (SDS) and height SDS The Secondary Objectives of the study are to assess the effect of 6-12 months treatment with nutritional supplementation standardized formula, in short and lean female adolescents on BMI SDS, growth velocity, time to puberty, quality of life and self-esteem The study will continue for 6 months of intervention versus active placebo, with additional optional 6 months (an extension period), in which participants at both groups, the intervention and the placebo, will be offered to continue their participation in the study with the study supplement. All analyses of the effect's on primary and secondary outcome measurements will take into account the consumption rate of the study formula/placebo

ELIGIBILITY:
Inclusion Criteria:

* Girls aged ≥9 years old
* Prepubertal - Tanner stage 1. (gonadarche) Breast at Tanner stage 1)
* Height and weight ≤ 10th percentile for age and gender.
* Height-SDS ≥ -2.5 SDS
* BMI-SDS>-2 SDS
* Low proportion between weight and height
* Signing inform consent forms

Exclusion Criteria:

* Diagnosis of Growth Hormone (GH) Deficiency or treatment with GH
* Any known chronic disease or dysmorphic syndrome including: bone diseases, organic brain diseases, neurological disease, past or current malignancy, chronic cardiac, renal or pulmonary problems
* Any known gastrointestinal disease including malabsorption
* Any known organic reason for growth retardation
* Any chronic treatment with medication that might affect appetite, weight or growth (for example SSRI's).

Ages: 9 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2015-06; Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Weight SDS (standard deviation score) | At 12 months
  Standard deviation score of patient's weight at 12 months
Height SDS (standard deviation score) | At 12 months
  Standard deviation score of patient's height at 12 months
Weight SDS (standard deviation score) | At 6 months
  Standard deviation score of patient's weight at 6 months
Height SDS (standard deviation score) | At 6 months
  Standard deviation score of patient's height at 6 months

SECONDARY OUTCOMES:
BMI SDS (standard deviation score) | At 12 months
  Standard deviation score of patient's BMI at 12 months
BMI SDS (standard deviation score) | At 6 months
  Standard deviation score of patient's BMI at 6 months
Growth velocity | At 12 months
  Growth velocity measured as delta height divided by 12 months
Growth velocity | At 6 months
  Growth velocity measured as delta height divided by 6 months
Quality of life Questionnaire | At 12 months
  Quality of life measured by quality of life questionnaire
Quality of life Questionnaire | At 6 months
  Quality of life measured by quality of life questionnaire
Self-esteem Questionnaire | At 12 months
Self-esteem Questionnaire | At 6 months

OTHER OUTCOMES:
Time to puberty initiation | At 12 months
  Duration of time until breast at tanner stage >=2
Sleep Assessment Questionnaire | At 6 months
Sleep Assessment Questionnaire | At 12 months
Physical Activity Questionnaire | At 6 months
Physical Activity Questionnaire | At 12 months
Study Participation Questionnaire | At 6 months
Study Participation Questionnaire | At 12 months
Family Eating and Activity Habits Questionnaire | At 6 months
Family Eating and Activity Habits Questionnaire | At 12 months
Parents Stands Towards Healty Lifestyle Questionnaire | At 12 months
Parents Stands Towards Healty Lifestyle Questionnaire | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, Prof, Principal Investigator — Schneider Children's Medical Center
Locations (3):
- Israel (3):
  - Soroka Medical Center, Beersheba
  - Schneider Children's Medical Center, Petah Tikva
  - Assaf Harofe, Rishon LeZiyyon